CLINICAL TRIAL: NCT04502095
Title: Does Prophylactic Antibiotic Decrease the Rate of Urinary Tract Infection After Robot Assisted Radical Cystectomy
Brief Title: Prophylactic Antibiotics for Urinary Tract Infections After Robot-Assisted Radical Cystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 573720; NCI-2020-04928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 573720 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-07-24; First posted 2020-08-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Bladder Carcinoma; Refractory Bladder Carcinoma; Urinary Tract Infection
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Tract Infections | interventions — Clindamycin; Ertapenem; Levofloxacin; Ofloxacin; Nitrofurantoin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (trimethoprim-sulfamethoxazole, nitrofurantoin) (Experimental): Patients receive ertapenem PO, levofloxacin PO, or clindamycin PO induction therapy per standard of care. At the time of full diet, patients receive trimethoprim-sulfamethoxazole PO daily or nitrofurantoin PO daily on days 1-30. Patients complete a drug diary for each day they receive the antibiotic.
  Interventions: Drug: Clindamycin; Other: Diary; Drug: Ertapenem; Drug: Levofloxacin; Drug: Nitrofurantoin; Drug: Trimethoprim-Sulfamethoxazole
- Group II (standard of care) (Active Comparator): Patients receive ertapenem PO, levofloxacin PO, or clindamycin PO induction therapy per standard of care.
  Interventions: Drug: Clindamycin; Drug: Ertapenem; Drug: Levofloxacin

INTERVENTIONS:
Drug: Clindamycin — Given PO
  Other Names: Cleocin
Other: Diary — Complete drug diary
  Arms: Group I (trimethoprim-sulfamethoxazole, nitrofurantoin)
Drug: Ertapenem — Given PO
Drug: Levofloxacin — Given PO
  Other Names: (S)-9-Fluoro-2,3-dihydro-3-methyl-10-(4-methyl-1-piperazinyl)-7-oxo-7H-pyrido(1,2,3-de)-1,4-benzoxazine-6-carboxylic Acid Hydrate (2:1); Levaquin; Levofloxacin Hydrate; Quixin
Drug: Nitrofurantoin — Given PO
  Other Names: Macrobid; Macrodantin
  Arms: Group I (trimethoprim-sulfamethoxazole, nitrofurantoin)
Drug: Trimethoprim-Sulfamethoxazole — Given PO
  Other Names: Bactrim; Bactrim DS; Bactrimel; Centran; Centrin; Co-Trimoxazole; Cotrim; Cotrimoxazole; Eslectin; Insozalin; Septra; SMZ-TMP; Sulfamethoprim; Sulfatrim; Sulmeprim; TMP-SMX; Trimedin; Trimezole; Uroplus
  Arms: Group I (trimethoprim-sulfamethoxazole, nitrofurantoin)

SUMMARY:
This trial investigates whether a one-month course of preventative (prophylactic) antibiotics helps to reduce urinary tract infections after robot-assisted surgery to remove all of the bladder as well as nearby tissues and organs (radical cystectomy). Urinary tract infections are a common occurrence after robot-assisted radical cystectomy. Antibiotics such as trimethoprim-sulfamethoxazole or nitrofurantoin may prevent or control infections in patients with urinary tract infection and may help improve their response to radical cystectomy. Information gained from this study may help researchers to predict patient complications and identify better ways to manage these complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the utilization of a prophylactic antibiotic during the postoperative period will decrease the rate of urinary tract infection (UTI) post robot-assisted radical cystectomy.

SECONDARY OBJECTIVE:

I. To identify pre- and post-operative factors that may be associated with the development of a 90-day UTI following radical cystectomy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (ANTIBIOTIC): Patients receive ertapenem Intravenously (IV), levofloxacin, or clindamycin IV at induction per standard of care. At the time of full diet, patients receive trimethoprim-sulfamethoxazole PO daily or nitrofurantoin PO daily on days 1-30. Patients complete a drug diary for each day they receive the antibiotic.

GROUP II (CONTROL): Patients receive ertapenem IV, levofloxacin IV or clindamycin IV at induction per standard of care.

After surgery, patients are followed up to 120 days.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that electively chooses to have a cystectomy is eligible to participate in the study. Indications for a person who may undergo a cystectomy include having a diagnosis of muscle-invasive bladder cancer (MIBC) or refractory non-muscle invasive bladder cancer (NMIBC)
* Any patient that will electively choose to have a robot-assisted radical cystectomy and is able to provide consent
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients with a history of myasthenia gravis
* Patients with a history of QT prolongation or taking other drugs that prolong corrected QTc (QTc) should be excluded
* Patients with renal dysfunction, creatinine clearance (mL/min) < 30
* Pregnant or nursing female participants
* Females who receive a fertile sex sparing robot-assisted radical cystectomy (RARC)
* Unwilling or unable to follow protocol requirements
* Patients who receive a prophylactic antibiotic or antibiotic for any other reason prior to discharge
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
90-day urinary tract infection (UTI) status | At 90 days after surgery
  Will be treated as dichotomous data and will be summarized by group using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Identify pre-operative factors associated with the development of UTI | Up to 120 days after surgery
  stratified logistic regression models (stratified by antibiotic use)
Development of Clostridium difficile (C Diff) | up to 120 days after surgery
  Will be evaluated in patients who received prophylactic antibiotics.
Infections occurring during antibiotic use | Up to 120 days after surgery
  To identify which antibiotic is better suited as a prophylactic, comparisons will be made using two-sided Mann-Whitney U and Fisher's exact tests for continuous and categorical variables, respectively.
Identify post operative factors associated with the development of UTI | Up to 120 days after surgery
  stratified logistic regression models (stratified by antibiotic use)

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid A Guru, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States